CLINICAL TRIAL: NCT03521609
Title: Emotional Intelligence in Patients With Addictive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-INT-2017-106
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Intelligence Intervention (Experimental): Patient's emotional abilities will be stimulated by means of a brief intervention in a group format (nine sessions). In these sessions we will use both projective and guided-fantasy techniques for the emotional diagnosis, as well as psychoeducational workshops of both emotional education and emotional intelligence development.
  Interventions: Behavioral: Emotional intelligence intervention

INTERVENTIONS:
Behavioral: Emotional intelligence intervention — Brief group intervention based on emotional intelligence

SUMMARY:
The study aims to evaluate the level of emotional intelligence in patients diagnosed with substance use disorder and to evaluate the benefits in emotional skills after a brief intervention based on emotional intelligence.

DETAILED DESCRIPTION:
Patients will be recruited by consecutive non-probabilistic sampling in the Addictions Day Hospital of the Addictions Unit of the Hospital de la Santa Creu i Sant Pau in Barcelona. The level of emotional intelligence will be assessed through the following measurement instruments: MSCEIT for the objective emotional intelligence coefficient and the TMMS-24 for the perceived emotional intelligence. Patients will attend 9 sessions of brief group intervention based on emotional intelligence and pre-post intervention differences in participants' TMMS-24 scores will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Substance Use Disorder (DSM-5)
* 18 to 80 years old

Exclusion Criteria:

* Presence of severe psychopathological alteration (including severe intoxication)
* Inability to understand the Spanish language or difficulties writing or reading

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in perceived emotional intelligence, measured with the Spanish version of the Trait Meta-Mood Scale (Fernandez-Berrocal, Extremera & Ramos, 2004). | Changes from baseline scores at 2-months scores
  The Trait Meta-Mood Scale (TMMS-24) is a 24-item self-report instrument with three subscales measuring three key aspects of perceived emotional intelligence: Attention, Clarity and Repair. Each of these three subscales consists of eight items with a 5-point Likert response format (ranging from 1 to 5). Subscale total scores are obtained by summing responses to all items and thus range from 8 to 40, with higher scores indicating greater level of the characteristic assessed.
Score on an ability measure of emotional intelligence, the Spanish version of the Mayer-Salovey-Caruso Emotional Intelligence Test (Extremera & Fernández-Berrocal, 2016). | Pre-intervention only
  The Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) consists of 141 items that yield an overall emotional intelligence (EI) score and two EI area scores: the Experiential EI and Strategic EI scores. The aforementioned scores have a mean of 100 and a standard deviation of 15, with higher scores indicating greater emotional intelligence.

SECONDARY OUTCOMES:
Change in self-esteem, measured with the Spanish version of the Rosenberg Self-Esteem Scale (Martin-Albo, Núñez, Navarro & Grijalvo, 2007). | Changes from baseline scores at 2-months scores
  The Rosenberg Self-Esteem Scale (RSES) is a self-report measure of global self-esteem. It consists of ten items with a 4-point Likert response format (ranging from 1 to 4). The RSES total score is obtained by summing responses to all items and thus ranges from 10 to 40, with higher scores indicating greater self-esteem.
Change in subjective happiness, measured with the Spanish version of the Subjective Happiness Scale (Extremera & Fernández-Berrocal, 2013). | Changes from baseline scores at 2-months scores
  The Subjective Happiness Scale (SHS) is a self-report measure of global subjective happiness. It consists of four items with a 7-point Likert response format (ranging from 1 to 7). The SHS total score is obtained by averaging responses to all items and thus ranges from 1 to 7, with higher scores indicating greater happiness.
Change in life satisfaction, measured with the Spanish version of the Satisfaction with Life Scale (Vásquez, Duque & Hervás, 2013). | Changes from baseline scores at 2-months scores
  The Satisfaction with Life Scale (SWLS) is a self-report measure of life satisfaction. It consists of five items with a 7-point Likert response format (ranging from 1 to 7). The SWLS total score is obtained by summing responses to all items and thus ranges from 5 to 35, with higher scores indicating greater life satisfaction.
Change in anxiety levels, measured with the Spanish version of the State-Trait Anxiety Inventory - State subscale (Spielberger, Gorsuch & Lushene, 2011). | Changes from baseline scores at 2-months scores
  The State-Trait Anxiety Inventory - State subscale (STAI-S) is a self-report measure of state anxiety. It consists of 20 items with a 4-point Likert response format (ranging from 0 to 3). The STAI-S total direct score is obtained by summing responses to all items and thus ranges from 0 to 60, with higher scores indicating greater levels of state anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Seyla De Francisco Prófumo, RN, Principal Investigator — Fundació de Gestió Snitària de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Santa Creu i Sant Pau Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided